CLINICAL TRIAL: NCT03710460
Title: Effect of the Administration of the Combination of Dapagliflozin Plus Metformin XR Versus Monotherapies on Anthropometric Indicators in Patients With Grade 1 Obesity.
Brief Title: Effect of Dapagliflozin/Metformin XR vs Monotherapies on Anthropometric Indicators in Obesity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Karina Griselda Pérez Rubio, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dapa-MetforminXR in Obesity
Record Dates: First submitted 2018-10-04; First posted 2018-10-18 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2022-06

CONDITIONS: Obesity
Keywords: Obesity; Dapagliflozin; Metformin XR; Visceral adiposity
MeSH Terms: conditions — Obesity | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dapagliflozin (Experimental): Dapagliflozin capsules, 10 mg, one per day before breakfast during 12 weeks.
  Interventions: Drug: Dapagliflozin
- Dapagliflozin plus metformin XR (Experimental): Dapagliflozin plus metformin XR capsules, 10/1000 mg, one per day before breakfast during 12 weeks.
  Interventions: Drug: Dapagliflozin plus Metformin XR
- Metformin XR (Experimental): Metformin XR capsules, 1000 mg, one per day before breakfast during 12 weeks.
  Interventions: Drug: Metformin XR

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg, one per day before breakfast during 12 weeks.
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Dapagliflozin plus Metformin XR — 10/1000 mg, one per day before breakfast during 12 weeks.
  Other Names: XigDuo
  Arms: Dapagliflozin plus metformin XR
Drug: Metformin XR — 1000 mg, one per day before breakfast during 12 weeks.
  Arms: Metformin XR

SUMMARY:
Obesity has increased to alarming levels in the world. Currently it is estimated that it occurs in a third of the world's population and it is expected that by 2030, 20% of the world's adult population will suffer from obesity and 38% will be overweight, and it is important to highlight that Mexico is among the first in obesity in adults and children.

Obesity leads to the development of diseases such as diabetes mellitus type 2, dyslipidemias, metabolic syndrome, heart problems, among others.

The treatment for obesity in the first instance are changes in lifestyle, changes in diet and exercise that have shown, in most patients, have little long-term adherence. There are also drugs that promote weight loss by modifying the appetite or absorption of macronutrients.

Dapagliflozin plus metformin XR is a medicine composed with an oral antidiabetic of the group of inhibitors of SGLT2 that has shown to have significant side effects in the weight reduction and visceral adiposity in people with obesity and in patients with diabetes mellitus type 2, it is also composed with metformin which also has effects on weight loss in people with and without type 2 diabetes mellitus.

For these reasons, evaluating this compound drug in people with obesity could provide high impact information as a complement for the treatment of this condition when compared to the effects produced by monotherapies.

DETAILED DESCRIPTION:
A double-blind, randomized clinical trial of three pharmacological groups in 33 patients with a diagnosis of grade 1 obesity in accordance with the World Health Organization (WHO) without treatment.

They will be assigned randomly three groups of 11 patients, each one will receive 10 mg of dapaglizflozin (Forxiga, Astra Zeneca), 1000 mg of metformin XR or 10/1000 mg of dapagliflozin plus metformin XR, one time per day before having break-fast during 12 weeks.

The body weight, body mass index (BMI), adiposity %, visceral adiposity, fat mass, lean mass, waist circunference,waist-hip index, arterial pressure, and laboratory parameters as a glucose, triglicerides, cholesterol, High density lipoprotein (c-HDL), low density lipoprotein (c-LDL), uric acid, creatinin, C reactive protein, adiponectin and interleukin 10, leptin and TNF-∝will be measures.

This protocol is already approved by the local ethics committee and written informed consent it's going to be obtained from all volunteers.

Statistical analysis will be presented through measures of central tendency and dispersion, average and deviation standard for quantitative variables; frequencies and percentages for variable qualitative. Qualitative variables will be analyzed by X2, will be used for differences inter-group Kruskal-Wallis Test and Wilcoxon Test for the within-groups differences. It will be considered statistical significance p ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed grade 1 obesity according to the WHO criteria:
* -Body Mass Index (BMI) between 30 to 34.9 kg/m²
* No pharmacological treatment for obesity
* Stable weight during the last 3 months

Exclusion Criteria:

* Pregnancy or breast-feeding
* History of kidney or liver disease
* Drugs or supplements consumption with proven properties that modify the behavior of obesity
* Total cholesterol >240 mg/dL
* Triglycerides >500mg/dL
* Glucose ≥126 mg/dL or HbA1C ≥6.5%.
* Patients who smoke daily for the last 6 months
* Hypersensitivity to dapagliflozin or metformin XR

Ages: 31 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Body Weight | Baseline to week 12
  The body weight will be measured at baseline to week 12 with a bioimpedance balance and the entered values reflect the body weight at week 12
Body Mass Index | Baseline to week 12
  Body Mas Index will be calculated at baseline to week 12 with the Quetelet index formula and the entered values reflect the body mass index at week 12
Adiposity percentage | Baseline, week 4, week 8 and week 12
  The adiposity percentage will be measured at baseline to week 12 with a bioimpedance balance and the entered values reflect the adiposity percentage at week 12
Visceral adiposity | Baseline to week 12
  Visceral adiposity will be measured at baseline to week 12 with a bioimpedance balance and the entered values reflect the visceral adiposity in square meter at week 12
Lean mass | Baseline to week 12
  The lean mass will be measured at baseline to week 12 with a bioimpedance balance and the entered values reflect the lean mass at week 12
Fat mass | Baseline to week 12
  The fat mass will be measured at baseline to week 12 with a bioimpedance balance and the entered values reflect the fat mass at week 12
Waist circumference | Baseline to week 12
  Waist circumference will be evaluated with the method proposed by ISAK.
Waist-hip ratio | Baseline to week 12
  The waist-hip ratio will be calculated as waist measurement divided by hip measurement

SECONDARY OUTCOMES:
Interleukin 10 levels IL-10 | Baseline and week 12
  Interleukin levels will be evaluated at baseline and week 12 by Enzyme-Linked ImmunoSorbent Assayed (ELISA) the entered values reflect the total interleukin 10 level at week 12
Adiponectin levels. | Baseline and week 12
  adiponectin levels will be evaluated at baseline and week 12 by Enzyme-Linked ImmunoSorben Assayed (ELISA) the entered values reflect the total adiponectin levels at week 12
C-reactive protein levels | Baseline and week 12
  C-reactive protein levels will be evaluated at baseline and week 12 by Enzyme-Linked ImmunoSorbent Assayed (ELISA) the entered values reflect the total C-reactive protein levels levels at week 12
Leptin levels | Baseline and week 12
  Leptin levels will be evaluated at baseline and week 12 by Enzyme-Linked ImmunoSorbent Assayed (ELISA) the entered values reflect the total leptin levels levels at week 12
TNF-α levels | Baseline and week 12
  Tumor necrosis factor alpha (TNF-α) levels will be evaluated at baseline and week 12 by Enzyme-Linked ImmunoSorbent Assayed (ELISA) the entered values reflect the total TNF-αl levels levels at week 12
Total cholesterol | Baseline to Week 12
  Total cholesterol levels will be evaluated at baseline and week 12 by enzymatic/colorimetric techniques and the entered values reflect the total cholesterol level at week 12
HDL cholesterol | Total high density lipoprotein cholesterol levels will be evaluated at baseline and week 12 by enzymatic/colorimetric techniques and the entered values reflect the high density lipoprotein cholesterol level at week 12
  High density lipoprotein cholesterol (HDL-C)
LDL cholesterol | Total low density lipoprotein cholesterol levels will be evaluated at baseline and week 12 by enzymatic/colorimetric techniques and the entered values reflect the low density lipoprotein cholesterol level at week 12
  Low density lipoprotein cholesterol (LDL-C)
Triglycerides levels | Baseline to Week 12
  Triglycerides levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the triglycerides level at week 12
Fasting glucose levels | Baseline to Week 12
  The fasting glucose levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at week 12.
Creatinine levels | Baseline to Week 12
  Creatinine levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques
Uric acid levels | Baseline to Week 12
  Uric acid levels will be evaluated at baseline and week 12 with enzymatic/colorimetric techniques
Systolic blood pressure | Baseline, week 4, week 8 and week 12
  blood pressure will be measured at baseline week 4, week 8 and week 12 with a digital sphygmomanometer. Values will be expressed in millimeters of mercury (mmHg).
Diastolic blood pressure | Baseline, week 4, week 8 and week 12
  blood pressure will be measured at baseline week 4, week 8 and week 12 with a digital sphygmomanometer. Values will be expressed in millimeters of mercury (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Gonzalez Ortiz, MD MSc Phd, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico